CLINICAL TRIAL: NCT05798013
Title: Effectiveness of Digital Health Management on Patients With Head and Neck Vascular Stenosis: A Multicenter, Cluster Randomized Controlled Trial Based on Chinese Population
Brief Title: Effectiveness of Digital Health Management on Patients With Head and Neck Vascular Stenosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ENHEARTEN
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Vascular Stenosis
Keywords: head and neck vascular stenosis; digital health management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital health management intervention Group (Experimental): Patients in the trial group receives intervention management from the digital health management platform, including reminding patients to take medication on time, monitoring and managing risk factors, reminding patients to have regular checkups and regular follow-ups, and pushing personalized science based on patients' risk factors, etc. Meanwhile, the platform's customer service staff regularly follows up with patients and reminds them of health management, and regularly invites experts to conduct formal medical science conferences for patients.
  Interventions: Behavioral: Digital health management
- Control group (No Intervention): The group doesn't not receive intervention reminders and customer service supervision from the platform, but receives the same follow-up visits.

INTERVENTIONS:
Behavioral: Digital health management — The digital health management platform mainly includes reminding patients to take medication on time, monitoring and managing risk factors, reminding patients of regular review and regular follow-up, pushing personalized science according to patients' risk factors, etc., as well as following up and supervising patients' health management, and conducting regular formal medical science conferences.
  Arms: Digital health management intervention Group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of digital health management for intervention on Chinese population with head and neck vascular stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria of the clusters

   Hospitals with the qualification of "head and neck ultrasound center" in China.
2. Inclusion criteria for individuals

   * (1)Age ≥ 35 years old, with no restriction on gender.
   * (2)Patients with clinically diagnosed head and neck stenosis or occlusion, including mild, moderate or severe stenosis or occlusion of the carotid artery and mild, moderate or severe stenosis or occlusion of the intracranial artery.
   * (3)Ability to use a smartphone and have a mobile application installed on the handset.
   * (4)Subjects or their legal representatives agreed to the study and signed the project informed consent form.

Exclusion Criteria:

1. Exclusion criteria for the clusters

   The included centers did not have the capacity to undertake the trial.
2. Exclusion criteria for individuals

   * (1)Combination of severe systemic diseases such as respiratory failure, renal failure, gastrointestinal bleeding, coagulation dysfunction, malignancy, etc.
   * (2)Patients with a life expectancy of less than 2 years or who are unable to complete the study for other reasons.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102072 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
New-onset stroke events at 24 months | 24 months
  New-onset stroke events include ischemic stroke, transient ischemic attack, and hemorrhagic stroke.

SECONDARY OUTCOMES:
New-onset stroke events at 12 months | 12 months
  New-onset stroke events include ischemic stroke, transient ischemic attack, and hemorrhagic stroke.
Composite and separate indicators of new clinical vascular events at 12 and 24 months | 12 months, 24 months
  Clinical vascular events included ischemic stroke, transient ischemic attack, hemorrhagic stroke, myocardial infarction, and vascular death.
All-cause deaths at 24 months | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China